CLINICAL TRIAL: NCT02832479
Title: Costs of Care and Adherence to Treatment for Cystic Fibrosis.
Acronym: COMURA MUCOBS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0698
Record Dates: First submitted 2016-06-21; First posted 2016-07-14 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evolution of medical care for patients with cystic fibrosis appeared in recent years: prolongation of life expectancy with consequently increased comorbidities and the use of lung transplantation, systematic neonatal screening of new born since 2002, prescription of expensive new molecules or new presentation. This evolution justifies to realize an update of statistics of costs of care and to assess adherence to treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis,
* Followed by one of the cystic fibrosis center of the Rhône-Alpes region (pediatric and adult of Lyon and Grenoble)
* Affiliated to the general scheme of health insurance,
* And domiciled in the Rhône-Alpes region.

Exclusion Criteria:

* Transplanted patients

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cystic fibrosis living in Rhône-Alpes region
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
treatment cost | 12 months

SECONDARY OUTCOMES:
adherence rate for chronic treatment | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices civils de Lyon, centre hospitalier lyon Sud, Pierre-Bénite, France